CLINICAL TRIAL: NCT03116386
Title: Reduced Time on Floor After Falls at Night of People Living in Long Term Care Facilities - NoDelayFall Study
Brief Title: Time Spent on Floor After Falls of Frailty People Overnight
Acronym: NoDelayFall
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability of the ETOLYA®'s manufacturer to furnish the promised functionalities as those which had to be recorded for assessment of the study's end points
Sponsor: Centre Hospitalier Annecy Genevois (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2016-A01799-42
Record Dates: First submitted 2017-04-06; First posted 2017-04-17 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2017-04

CONDITIONS: Dependence; Fall From Bed; Fall Injury; Fall in Nursing Home; Cognition Disorders
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Intervention Model Description: Run-in period then 6 months control period and then 6 months experimental period with activation of all the functions of Etolya-F® (the device used in the study)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- run-in period (Other): In order to improve the precision of data, the run-in period is dedicated to sensitize the caregivers about the importance of
  * reporting all the falls occurring during the night
  * tracking in each resident's file, all informations about the estimate length of time spent on floor after a fall occurring during the night
  * and also reporting every other events occuring at night as wandering. All the beds will progressively equipped with the Etolya-F ® devices but the Etolya-F ® ddevices will stay off.
  Interventions: Other: run-in period
- control period (Sham Comparator): We expect 30 falls will occurr at night during this 6 months period. Etolya-F ® devices will be installed on the bed of all participant residents but with limited fonctionnalities i.e. only the length of absence in the bed will be recorded (difference between time of detection of the beginning of absence in the bed and time where the resident will be found by the caregivers out of his bed).
  Interventions: Device: Control period
- Etolya-F ® devices (Experimental): We also expect 30 falls will occur at night during this 6-month period. Etolya-F ® devices will be used with all their functionalities i.e. permit detection of absence in the bed, activation of a lighting environment when the resident gets up from his bed, transmission of alert to caregivers through the centralized system of sick call if the resident do not return to bed after 15 minutes and recording the time when caregivers will find the resident out of bed, distinguishing between a fall and a night wandering in the room or corridors without a fall
  Interventions: Device: Etolya-F ® devices

INTERVENTIONS:
Other: run-in period — observational time i.e. baseline situation
  Arms: run-in period
Device: Control period — neither activation of any lighting environment when the resident gets up from his bed nor alert if the resident did not return to bed after 15 minutes Etolya-F ® devices will only permit detection and recording of the moment of the elderlly will leave his/her bed and recording of the moment the elderly will be found by caregivers
  Arms: control period
Device: Etolya-F ® devices — Etolya-F ® devices will permit detection of absence in the bed, activation of a lighting environment when the resident gets up from his bed, transmission of alert to caregivers through the centralized system of sick call if the resident do not return to bed after 15 minutes and recording the time when caregivers will find the resident out of bed, distinguishing between a fall and a night wandering in the room or corridors without a fall
  Arms: Etolya-F ® devices

SUMMARY:
In the context of reduce staff for supervision of dependent elderly, automated risk alert systems could have a positive impact on the organization of night care by better targeting monitoring. Residents' sleep could be less affected with use of automatic alert system than by systematic monitoring visits. One study shows an improvement in the humor of residents after the use of such a system.

The hypothesis of the study is that the use of a bed-raising detection system linked with the activation of a lighting environment and a caregivers alert system (Etolya-F® gerontechnology device, Anaxi Technology Company) would reduce intervention time in this population, thus limiting the time spent on floor and its physical and psychological consequences.

DETAILED DESCRIPTION:
In France in 2011, more than 575000 elderly lived in long term care facilities. Most of them had comorbidities.

The most frequent reason for admitting in long term care facilities is the worsening of health status of elderly, often triggered by a fall. Elderly living in long term care facilities have frequently several comorbidities; the first ones are Alzheimer and related diseases. The proportion of such very dependent institutionalized people has risen for the last recent years and they represent a population at very high risk of falling. In an epidemiological analysis of more than 70,000 falls from residents of Bavarian nursing homes, the prevalence of fall was estimated at 1.49 falls for women and 2.18 for men. Those results didn't take into account the fact that people could fall more than once a day. In Alzheimer people (or people with related diseases) who lived in long term care facilities, the incidence of falls was even highest with 2.7 falls per resident per year.

The consequences of falls are not only physical injuries (wounds, fractures); they are frequently associated with psychological repercussions as loss of self-confidence, fear of new falls, reduction of abilities of moving which lead into declining of daily activities and loss of autonomy.

The incapacity of getting up alone is reported by more than a third of patients who have fallen, even if the fall is not complicated by a fracture. The length of time people stay on floor is directly link to the ability of the elderly person to give an alarm and to the presence or not of someone else to help him/her to get up. Patients who live in long term care facilities have limited functional capabilities not compatible with an operational use of active alarm systems.

In long term care facilities, 30-40% of falls occur between 8pm and 8am. Falls occurring at night seem to be associated with more severe injuries. Staff are less numerous at night with only 3 to 4 caregivers for 100 people.

To the best of the knowledge of the investigators, delay intervention time after a fall occurring at night has never been studied. Based on the investigators' experience, elderly people can only be discovered and helped when caregivers find them on floor on the occasion of a planned surveillance visit. These visits are carried out every 2 to 4 hours at night.

Automated alarms are used to alert staff to situations where there is a high risk of falling: an attempt to lift an armchair from a person who cannot stand or to detect the night-time rise of a high-risk people with the use of various sensors (pressure sensors connected to the mattress or environmental sensors).

In the context of staff reduced at night for the supervision of dependent elderly, automated risk alert systems could also have a positive impact on the organization of night care by better targeting monitoring. Residents' sleep could be less affected with use of automatic alert system than by systematic monitoring visits. One study shows an improvement in the humor of residents after the use of such a system.

The hypothesis of the study is that the use of a bed-raising detection system linked with the activation of a lighting environment and a personnel alert system (Etolya-F® gerontechnology device, Anaxi Technology Company) would reduce intervention time in this population, thus limiting the time spent on floor and its physical and psychological consequences.

ELIGIBILITY:
Inclusion Criteria:

* elderly people who are resident in long term care facilities
* non opposed to participate to the study or whose his/her legal representative is not opposed to the participation of the resident to the study

Exclusion Criteria:

* the resident's bed can not be equipped with the ETOLYA-F® device for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Time for caregivers to find a resident who falls at night, before and after use of the Etolya-F® device | 2 periods of 6 months
  Delay elapsing between the moment a resident has left his/her bed and the time he/she was found by caregivers, on floor after a fall at night

SECONDARY OUTCOMES:
Diagnostic performance of the Etolya-F® device in the detection of night falls | 2 periods of 6 months
  sensitivity and specificity of Etolya-F®
Traumatic consequences of falls | 2 periods of 6 months
  Number of night falls resulting in hospitalization, fracture (s) or wound (s) requiring suture (s) or death

OTHER OUTCOMES:
Number of night falls | 2 periods of 6 months
  Number of actual falls occurring at night during each of the two study periods
Number of night wandering | 2 periods of 6 months
  Number of actual wandering occurring at night during each of the two study periods

CONTACTS AND LOCATIONS:
Overall Officials: Dr Matthieu DEBRAY, MD, Study Director — CH Annecy Genevois; Dr Nathalie RUEL, MD, Principal Investigator — CH Annecy Genevois
Locations (1):
- Résidence St François CH ANNECY-GENEVOIS, Annecy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rapp K, Becker C, Cameron ID, Konig HH, Buchele G. Epidemiology of falls in residential aged care: analysis of more than 70,000 falls from residents of bavarian nursing homes. J Am Med Dir Assoc. 2012 Feb;13(2):187.e1-6. doi: 10.1016/j.jamda.2011.06.011. Epub 2011 Aug 4. PMID 21816682
- [Background] Pellfolk T, Gustafsson T, Gustafson Y, Karlsson S. Risk factors for falls among residents with dementia living in group dwellings. Int Psychogeriatr. 2009 Feb;21(1):187-94. doi: 10.1017/S1041610208007837. Epub 2008 Oct 6. PMID 18834557
- [Background] Jensen J, Lundin-Olsson L, Nyberg L, Gustafson Y. Falls among frail older people in residential care. Scand J Public Health. 2002;30(1):54-61. PMID 11928835
- [Background] Vu MQ, Weintraub N, Rubenstein LZ. Falls in the nursing home: are they preventable? J Am Med Dir Assoc. 2006 Mar;7(3 Suppl):S53-8, 52. doi: 10.1016/j.jamda.2005.12.016. PMID 16500282
- [Background] Lach HW, Parsons JL. Impact of fear of falling in long term care: an integrative review. J Am Med Dir Assoc. 2013 Aug;14(8):573-7. doi: 10.1016/j.jamda.2013.02.019. Epub 2013 Apr 16. PMID 23602257
- [Background] Fleming J, Brayne C; Cambridge City over-75s Cohort (CC75C) study collaboration. Inability to get up after falling, subsequent time on floor, and summoning help: prospective cohort study in people over 90. BMJ. 2008 Nov 17;337:a2227. doi: 10.1136/bmj.a2227. PMID 19015185
- [Background] Bergland A, Laake K. Concurrent and predictive validity of "getting up from lying on the floor". Aging Clin Exp Res. 2005 Jun;17(3):181-5. doi: 10.1007/BF03324594. PMID 16110729
- [Background] Lester P, Haq M, Vadnerkar A, Feuerman M. Falls in the nursing home setting: does time matter? J Am Med Dir Assoc. 2008 Nov;9(9):684-6. doi: 10.1016/j.jamda.2008.06.007. Epub 2008 Sep 25. PMID 18992702
- [Background] Pelissier C, Vohito M, Fort E, Sellier B, Agard JP, Fontana L, Charbotel B. Risk factors for work-related stress and subjective hardship in health-care staff in nursing homes for the elderly: A cross-sectional study. J Occup Health. 2015;57(3):285-96. doi: 10.1539/joh.14-0090-OA. Epub 2015 Apr 10. PMID 25864937
- [Background] Capezuti E, Brush BL, Lane S, Rabinowitz HU, Secic M. Bed-exit alarm effectiveness. Arch Gerontol Geriatr. 2009 Jul-Aug;49(1):27-31. doi: 10.1016/j.archger.2008.04.007. Epub 2008 Jun 3. PMID 18508138
- [Background] Banerjee S, Steenkeste F, Couturier P, Debray M, Franco A. Telesurveillance of elderly patients by use of passive infra-red sensors in a 'smart' room. J Telemed Telecare. 2003;9(1):23-9. doi: 10.1258/135763303321159657. PMID 12641889
- [Background] Lipsitz LA, Tchalla AE, Iloputaife I, Gagnon M, Dole K, Su ZZ, Klickstein L. Evaluation of an Automated Falls Detection Device in Nursing Home Residents. J Am Geriatr Soc. 2016 Feb;64(2):365-8. doi: 10.1111/jgs.13708. Epub 2016 Jan 19. PMID 26783046
- [Background] Tinetti ME, Williams CS. Falls, injuries due to falls, and the risk of admission to a nursing home. N Engl J Med. 1997 Oct 30;337(18):1279-84. doi: 10.1056/NEJM199710303371806. PMID 9345078
- [Background] Parker MJ, Gillespie WJ, Gillespie LD. Effectiveness of hip protectors for preventing hip fractures in elderly people: systematic review. BMJ. 2006 Mar 11;332(7541):571-4. doi: 10.1136/bmj.38753.375324.7C. Epub 2006 Mar 2. PMID 16513687
- See also: New technologies likely to improve gerontological practices and the daily life of elderly patients and their families — http://www.ladocumentationfrancaise.fr/var/storage/rapports-publics/074000390.pdf